CLINICAL TRIAL: NCT05493059
Title: Study of Cases of Cutaneous Leishmaniasis Treated With Miltefosine in French Guiana, Retrospective Study Before Clinical Trial (MILT 2022)
Brief Title: Study of Cases of Cutaneous Leishmaniasis Treated With Miltefosine in French Guiana, Retrospective Study
Acronym: MILT2022
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_028
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Cutaneous Leishmaniases; Treatment Adherence; Primary Health Care; Drug Evaluation
Keywords: Pentamidine; Amphotericin B; Meglumine Antimoniate; oral administration; intraveinous administration; intramuscular administration; French Guiana
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Treatment Adherence and Compliance | interventions — Data Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: * Mucocutaneous Leishmaniasis proven by culture and/or polymerase chain reaction (PCR)
  * Seen in French Guiana between 01/01/2017 and 01/04/2022, in dispensaries (CDPS) or in the Dermatology Department of the CHC
  * Having received treatment with Miltefosine
  * Patient who consented to participate in the study
  * Age equal or superior to 18 years
  Interventions: Other: Data collection; Other: Questionnaires

INTERVENTIONS:
Other: Data collection — o Retrospective data collection in database from medical records (clinical, parasitological and therapeutic data)
Other: Questionnaires — o Administration of two standardized questionnaires by telephone in prospective:
  * Dermatology Life Quality Index (DLQI)
  * Treatment Satisfaction Questionnaire for Medication (TSQM)

SUMMARY:
Miltefosine is the only oral treatment currently available for Cutaneous Leishmaniasis.

Despite several reports of good efficiency in other countries of South America, miltefosine remains limited to a compassionate use in France. The objective of this study is to collect data regarding the efficacy, safety and acceptability of miltefosine in patients treated in French Guiana since 2017.

DETAILED DESCRIPTION:
In French Guiana, Cutaneous Leishmaniasis is mostly caused by Leishmania guyanensis (80% of cases), followed by L. braziliensis (10%) and rarer species. L. guyanensis is usually treated with a single injection of pentamidine. However, pentamidine-resistant infections (10%) and all L. braziliensis are treated with either amphotericine B or meglumine antimoniate. These treatments can only be used during an hospitalization, which is the source of important indirect costs and discomforts for patients from the remote areas of French Guiana. Miltefosine is the only oral treatment available for Cutaneous Leishmaniasis. While it is widely used in South America (with good reported efficacy), the data available in France are scarce. This treatment, if available on a larger scale in France, would allow a treatment without hospitalization, which would be very suitable for French Guianese patients.

Our objective is to collect data on patients already treated with miltefosine in French Guiana (current indications being failure, side effect or impossible delivery of amphotericine B and meglumine antimoniate) in order to assess its efficacy, safety and acceptability. Patients treated with miltefosine at the Cayenne Hospital Center between 2017 and 2022 will be contacted by phone so as to answer questions regarding their quality of life during the infection and their satisfaction concerning miltefosine as a treatment. Data on their symptoms and general informations will be extracted from the medical files.

Primary objective: To assess the efficacy, tolerance and acceptability of Miltefosine among patients already treated with this drug as part of its AAC in French Guiana.

Observational, retrospective and prospective, monocentric study Research Involving Human Person Category 3 (RIPH3) - Non-Interventional (RNI) - Questionnaire (Jardé Law)

ELIGIBILITY:
Inclusion Criteria:

* Mucocutaneous Leishmaniasis proven by culture and/or polymerase chain reaction (PCR)
* Seen in French Guiana between 01/01/2017 and 01/04/2022, in dispensaries (CDPS) or in the Dermatology Department of the CHC
* Having received treatment with Miltefosine
* Patient who consented to participate in the study
* Age equal or superior to 18 years

Exclusion Criteria:

* Clinically suspected but not parasitologically proven leishmaniasis
* Refusal to participate
* Age < 18
* Patient under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting Mucocutaneous Leishmaniasis proven by culture and/or polymerase chain reaction (PCR) seen in French Guiana between 01/01/2017 and 01/04/2022, in dispensaries (CDPS) or in the Dermatology Department of the CHC and having received treatment with Miltefosine
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-08 (Estimated); Primary Completion 2022-08-08 (Estimated); Study Completion 2022-10-08 (Estimated)

PRIMARY OUTCOMES:
Disappearance of any lesion without the appearance of a new lesion, 6 months from the start of treatment with miltefosine | baseline
  The primary endpoint will be therapeutic success, defined as the disappearance of any lesion without the appearance of a new lesion, 6 months from the start of treatment with miltefosine.

SECONDARY OUTCOMES:
Proportion of treatment-emergent adverse events occurring during treatment | baseline
  Proportion of treatment-emergent adverse events occurring during treatment, categorized as follows: non-symptomatic laboratory abnormalities (mild); symptoms not leading to discontinuation or modification of treatment (moderate intensity); symptoms leading to discontinuation or dose reduction (severe intensity)
Patients' acceptability of treatment assessed after completion of treatment | baseline
  Patients' acceptability of treatment assessed after completion of treatment, by Treatment Satisfaction Questionnaire for Medication (TSQM) administered by telephone
Impact of Cutaneous Leishmaniasis on quality of life | baseline
  Impact of Cutaneous Leishmaniasis on quality of life, assessed retrospectively by Dermatology Life Quality Index (DLQI) questionnaire administered by telephone

CONTACTS AND LOCATIONS:
Overall Officials: Romain BLAIZOT, Principal Investigator — Centre Hospitalier de Cayenne, Dermatology